CLINICAL TRIAL: NCT02820025
Title: To Investigate the Effect and Mechanism of Respiratory Stimulant Doxapram on Facilitating Emergence From General Anesthesia Undergoing Elective Lumbar Surgery
Brief Title: The Effect and Mechanism of Respiratory Stimulant Doxapram on Facilitating Emergence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: mzk2015orexin
Record Dates: First submitted 2016-05-25; First posted 2016-06-30 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Doxapram; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- doxapram group (Experimental): the doxapram group iv doxapram 1mg/kg,
  Interventions: Drug: doxapram
- Controlled group (Placebo Comparator): the controlled group given equal volume of saline with the doxapram group.
  Interventions: Other: saline

INTERVENTIONS:
Drug: doxapram
  Arms: doxapram group
Other: saline
  Arms: Controlled group

SUMMARY:
The current study is designed to investigate the difference of plasma orexin A levels between doxapram group and controlled group at emergence time from sevoflurane-remifentanil anesthesia who will undergo elective lumbar surgery.

DETAILED DESCRIPTION:
BACKGROUND: General anesthesia has been widely used in clinics, while its mechanism is not fully clear.Delayed emergence from general anesthesia happens from time to time, which increases the occurrence of complications and economic burden of patients. The analeptics currently used in clinic have some side effects. Recently,studies have shown that orexin can facilitate emergence from general anesthesia.Because of its complex chemical structure and difficulty of synthetic process, a mountain of works needs to be done before its use in clinic. Doxapram has been widely used as a respiratory stimulant on patients. Recently the investigators found in patient that intravenous injection of doxapram would shorten the emergence time from general anesthesia, while its associated mechanism is unclear. Based on our previous discovery that injection of doxapram in patients could increase the plasma level of orexin - A, the investigators hypothesized that doxapram probably facilitate emergence from general anesthesia by promoting the release of orexin.

DESIGNING: Forty patients with ASA physical status I or II scheduled for elective lumbar surgery under general anesthesia (lasting for 2h to 4h) were enrolled. Anesthesia was induced with propofol 1-2mg/kg and sufentanyl 0.2-0.3μg/kg. Following muscle relaxation with iv cisatracurium besylate 0.2mg/kg endotracheal intubation was performed. Anesthesia was maintained with sevoflurane (inhalational concentration: 0.8-2.0 MAC) and target controlled infusion remifentanil (targeted concentration:2-6ng/ml ) along with an oxygen/air mixture (FiO2 =0.5). Muscle relaxation was maintained with intermittent. Inhalational concentration of sevoflurane and injected target concentration were titrated to maintain the bispectral index (BIS) between 40 and 60 during anesthesia. The end-tidal carbon dioxide level was maintained between 30 and 40 mmHg by controlled mechanical ventilation. When the surgery was completed the investigators adjust the concentration sevoflurane to 0.8MAC of the patient and targeted concentration of remifentanil to 2ng/ml then stop all anesthetics and adjust the oxygen flow to 6.0 L/min, at the same time the doxapram group iv doxapram 1mg/kg, the controlled group given equal volume of saline. Record time from stopping anesthetics to emergence. Arterial blood (2ml) was collected at the following time,such as before and 1h after induction of anesthesia, at emergence (1 min after tracheal extubation) and half an hour after tracheal extubation. This was centrifuged at 3000 rpm for 15min at -4 ◦C in order to separate plasma then stored at -80 ◦C until assay for orexin A concentrations.

EXPECTED RESULTS: The plasma orexin A of the doxapram group will be higher with the emergence time shorter than the controlled group.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is Adult (≥18 years old and ≤75 years old)
2. Participants with a Body Mass Index (BMI) 20-25 kg/m2
3. Participants with ASA physical status Ⅰor Ⅱ
4. Participants with Heart function rating Ⅰor Ⅱ
5. patients will undergo elective lumbar surgery and general anesthesia
6. The operation time is 2h to 4h.

Exclusion Criteria:

1. Participant is a pregnant woman or a nursing mother.
2. Participants have a history of narcotics allergic reactions.
3. indices of liver or kidney function is twice higher than normal.
4. Participants have a history or diagnosis of depression.
5. Participants have a history of Brain Trauma.
6. Participants have a history of narcotics addiction or drug addiction.
7. Participants or his family have an International Classification of Sleep Disorders diagnosis of obstructive sleep apnea syndrome.
8. patients are refuse this trail or are not able to sign informed consent. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
orexin A concentrations | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Wang, M.D., Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- Anesthesiology department of General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: Undecided